CLINICAL TRIAL: NCT02666014
Title: Comparison of Sugammadex Versus Neostigmine in Women at High Risk of Postoperative Nausea and Vomiting After Laparoscopic Gynaecological Surgery: A Randomized Controlled Trial
Brief Title: Sugammadex Versus Neostigmine for Postoperative Nausea and Vomiting After Laparoscopic Gynaecological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Principal Investigator, Deepak Mathur, Consultant Anaesthetist, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHF/FG581S/2013; SHF/FG581S/2013 (Other Grant/Funding Number: SingHealth Foundation Grant)
Record Dates: First submitted 2015-02-02; First posted 2016-01-28 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; nausea; vomiting; sugammadex; neostigmine
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex group (Active Comparator): Sugammadex 2 mg/Kg will be administrated as a single dose via intravenous injection upon completion of surgery and guided by peripheral nerve stimulation.
  The drug is to be diluted with normal saline to make up to 5 ml volume to maintain blinding.
  Interventions: Drug: Sugammadex
- Neostigmine group (Active Comparator): Neostigmine 0.040 mg/Kg, along with Atropine 0.015 mg/kg, diluted in normal saline to make up 5 ml total volume to maintain blinding.
  Neostigmine 0.040 mg/Kg, along with Atropine 0.015 mg/kg will be administrated as a single dose via intravenous injection upon completion of surgery and guided by peripheral nerve stimulation for reversal of neuromuscular blockade produced during surgery.
  Atropine sulfate-diphenoxylate hydrochloride combination will be an adjuvant drug to balance muscarinic side effects of Neostigmine, when Neostigmine is administered.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Reversal of neuromuscular blockade
  Other Names: Bridion
  Arms: Sugammadex group
Drug: Neostigmine — Reversal of neuromuscular blockade
  Arms: Neostigmine group

SUMMARY:
The laparoscopic technique is commonly employed for abdominal gynaecological surgery in women. Postoperative nausea and vomiting (PONV) may occur in 30% of women undergoing gynaecological surgery. In patients with multiple risk factors for nausea and vomiting, the incidence is up to 80%. PONV has a significant negative effect on patient satisfaction after anesthesia and is one of the most common causes for unexpected hospital admissions in day-surgery.

Sugammadex and Neostigmine are both drugs that are used to reverse the effect of muscle relaxation producing drugs that are commonly used during surgery. Neostigmine has been the drug of common use for this purpose, but PONV is reported with its usage.

With this research we intend to determine whether the trial drug Sugammadex would reduce the incidence of PONV in high-risk women after undergoing laparoscopic gynaecological surgery when compared to Neostigmine.

DETAILED DESCRIPTION:
More than 1500 laparoscopic abdominal gynaecological surgeries are performed at our Hospital every year and hence there is a need to provide excellent analgesia and minimize side effects from medications to improve patient satisfaction and outcomes. Postoperative nausea and vomiting (PONV) may occur in 30% of women undergoing gynaecological surgery. In a patient population with multiple risk factors (e.g. female gender, duration of surgery > 2 hours, non-smoker, history of PONV or a history of motion sickness), the incidence is up to 80%. PONV has a significant negative effect on patient satisfaction after anesthesia and is one of the most common causes for unexpected hospital admissions in day-surgery.

The primary aim of our study is to determine whether Sugammadex would reduce the incidence of self-reported postoperative nausea after surgery in high-risk women 24-hours after undergoing laparoscopic gynaecological surgery, when compared to Neostigmine. The secondary aims are to investigate the effects of Sugammadex on the severity of self-reported PONV at 6-hour; the quality of recovery score at 24-hours; total number of patients with PONV, pain intensity and overall satisfaction score with anaesthesia following laparoscopic gynaecological surgery in high-risk women. This study is intended as a double-blinded, randomised, single-center trial at KK Women's and Children's Hospital.

Sugammadex is a selective relaxant-binding agent that provides rapid reversal from neuromuscular blockade induced during general anaesthesia to facilitate surgical procedures. The main advantage of sugammadex is that its action is not dependent on inhibition of acetylcholinesterase when compared to traditional reversal agents such as Neostigmine. Therefore, sugammadex is not associated with the cholinergic side effects like nausea, vomiting and bradycardia. This present study intends to provide a new, effective anaesthetic regimen producing a reduction in side effects from surgery and anaesthesia, with higher patient satisfaction.

Sugammadex was identified as the first selective relaxant-binding agent providing rapid reversal from neuromuscular blockade induced during general anaesthesia when used to facilitate surgical procedures (Welliver 2006). The mechanism of Sugammadex differs from that of other commonly used reversal agents, such as neostigmine and edrophonium, which are reversible acetylcholinesterase inhibitors.

Neostigmine relies on inhibition of acetylcholinesterase, causing autonomic instability and side effect like headache, blurred vision, slowing of the heart rate (bradycardia), and gastrointestial symptoms including anorexia, nausea, vomiting, abdominal cramps and diarrhea. Hence, an anticholinergic drug such as atropine has to be administered concurrently to prevent excessive muscarinic effects such as bradycardia (Gilman 1980). A previous study (Lovstad et al 2001) showed that neostigmine increases the incidence of postoperative nausea and vomiting after gynaecological surgery compared to a placebo. However, in the current practice of providing neuromuscular blockade for laparoscopic surgery, maintenance of neuromuscular blockade is required to facilitate surgery, thereby making reversal agents necessary to prevent postoperative residual neuromuscular blockade.

Knowledge Gap:

Without preventative treatment, about 30% of patients undergoing general anaesthesia are likely to suffer postoperative nausea and vomiting (PONV) (Cohen et al, 1994; Apfel et al, 1999). In a patient population with multiple risk factors (e.g. female gender, duration of surgery > 2 hours, non-smoker, history of PONV or history of motion sickness), the incidence is up to 80%. PONV has a significant negative effect on patient satisfaction after anaesthesia and is one of the most common causes for unexpected hospital admissions after day-surgery.

Since at our Hospital more than 1500 laparoscopic gynaecological surgeries are performed every year, this a significant clinical problem. Unplanned hospital admissions due to postoperative nausea and vomiting after a low-risk, day-surgical, gynaecological procedure at our hospital accounted for 29 cases out of a total of 163 cases last year (18%). In fact, the Ministry of Health tracks unplanned hospital admission as a performance indicator.

Sugammadex is more expensive when compared to neostigmine, and therefore its use should be limited to the high-risk PONV group, in order to maximize its cost-benefit potential. Sugammadex was first approved for use in the European Union in 2008 and is also approved in Australia, Iceland, New Zealand and Norway. A recently published Cochrane systematic review on Sugammadex (Abrishami et al 2012) examined the efficacy and safety of Sugammadex and the authors concluded that Sugammadex was shown to be more effective than placebo (no medication) or neostigmine in reversing muscle relaxation caused by neuromuscular blockade during surgery and is relatively safe. Inadequate reversal of neuromuscular blockade may lead to breathing problems or hypoxia due to an inability to breathe adequately, potentially leading to prolonged hospitalisation, thereby causing increased healthcare costs.

Train-of-four (TOF) monitoring enables the anaesthetist to assess if neuromuscular blockade could be safely reversed. The expert recommendation is to reverse neuromuscular blockade when TOF is at least 2 (0 to 4, 0= dense neuromuscular blockade, 4= minimal neuromuscular blockade). Sugammadex may potentially lead to greater patient safety in anaesthesia and at the same time offer greater patient satisfaction in terms of reducing the side effects of neostigmine like nausea and vomiting. However, there is little evidence about the clinical outcomes after administration of Sugammadex, such as the incidence and severity of PONV after surgery and the quality of recovery and pain intensity in high-risk women following laparoscopic gynaecological surgery.

Our current proposal will compare Sugammadex with neostigmine in women at high-risk of PONV after laparoscopic gynaecological surgery. As this study is the first clinical trial targeting the population at high-risk of developing PONV and may change routine clinical practice. If our hypothesis is true, Sugammadex will provide a new anaesthetic regime with better patient safety and efficacy such as reduction in unplanned hospital admissions; reduction in anaesthetic complications such as nausea, vomiting and inadequate reversal of neuromuscular blockade routinely produced during anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Females
2. In-patients
3. Age ≥ 21 years
4. ASA class 1 or 2
5. Undergoing elective laparoscopic, abdominal, gynaecological surgery.
6. Weight ≥ 40 Kg or ≤ 100 Kg
7. At least 3 risk factors for nausea and vomiting
8. Able to give valid, informed consent
9. Duration of surgery expected to be 120 minutes or more.

Exclusion Criteria:

1. Less than 3 risk factors for PONV
2. Nausea and/or vomiting in the last 72-hours prior to surgery
3. Regular antiemetic or opioid use
4. Obesity, with body weight ≥ 100.1 Kg
5. History of drug or alcohol abuse
6. ASA III or worse
7. Laparoscopic surgery that is converted to open surgery
8. Age ≤ 20-years of age
9. Patients with unknown pregnancy status in pre-menopausal women or those currently pregnant or breast-feeding.
10. Smokers
11. Anaphylaxis or hypersensitivity to study drug(s)
12. Day surgery procedure, unsuitable for follow up at 6 and 24-hours postoperatively.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of self-reported, postoperative nausea at 24-hours | 24 hours after surgery
  Incidence of self-reported, postoperative nausea at 24-hours after neuromuscular blockade reversal with sugammadex or neostigmine, in women at high-risk of PONV, after undergoing laparoscopic gynaecological surgery.

SECONDARY OUTCOMES:
Incidence of self-reported PONV following administration of Sugammadex or Neostigmine reversal for neuromuscular blockade at 6-hours | 6 hours after surgery
  Incidence of self-reported PONV following administration of Sugammadex or Neostigmine reversal for neuromuscular blockade 6-hours following laparoscopic gynaecological surgery in women at high-risk of PONV.
Severity of self-reported PONV after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal at 6-hours and 24-hours | 6 and 24 hours after surgery
  Severity of self-reported PONV after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal at 6-hours and 24-hours after undergoing laparoscopic gynaecological surgery in women at high-risk of PONV.
total number of patients with PONV following laparoscopic gynaecological surgery. | up to 24 hours after surgery
  total number of patients with PONV
Pain intensity after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal in women at high-risk for PONV at 6- and 24-hours | 6 hours and 24 hours after surgery
  Pain intensity after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal in women at high-risk for PONV at 6-hours and 24-hours following laparoscopic gynaecological surgery.
Quality of recovery score after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal in women at high-risk of PONV at 24 hours | 24 hours after surgery
  Quality of recovery score after administration of Sugammadex or Neostigmine for neuromuscular blockade reversal in women at high-risk of PONV at 24 hours following laparoscopic gynaecological surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Sia, Study Chair — CMB, KK Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007362. doi: 10.1002/14651858.CD007362.pub2. PMID 19821409
- [Background] Lovstad RZ, Thagaard KS, Berner NS, Raeder JC. Neostigmine 50 microg kg(-1) with glycopyrrolate increases postoperative nausea in women after laparoscopic gynaecological surgery. Acta Anaesthesiol Scand. 2001 Apr;45(4):495-500. doi: 10.1034/j.1399-6576.2001.045004495.x. PMID 11300390
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Cohen MM, Duncan PG, DeBoer DP, Tweed WA. The postoperative interview: assessing risk factors for nausea and vomiting. Anesth Analg. 1994 Jan;78(1):7-16. doi: 10.1213/00000539-199401000-00004. PMID 8267183
- [Background] Dahl V, Pendeville PE, Hollmann MW, Heier T, Abels EA, Blobner M. Safety and efficacy of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in cardiac patients undergoing noncardiac surgery. Eur J Anaesthesiol. 2009 Oct;26(10):874-84. doi: 10.1097/EJA.0b013e32832c605b. PMID 19455040
- [Background] Miller RD. Sugammadex: an opportunity to change the practice of anesthesiology? Anesth Analg. 2007 Mar;104(3):477-8. doi: 10.1213/01.ane.0000255645.64583.e8. No abstract available. PMID 17312188
- [Background] Naguib M. Sugammadex: another milestone in clinical neuromuscular pharmacology. Anesth Analg. 2007 Mar;104(3):575-81. doi: 10.1213/01.ane.0000244594.63318.fc. PMID 17312211
- [Background] Yang LP, Keam SJ. Sugammadex: a review of its use in anaesthetic practice. Drugs. 2009;69(7):919-42. doi: 10.2165/00003495-200969070-00008. PMID 19441874